CLINICAL TRIAL: NCT03889691
Title: Does Watching Video Increase the Perioperative Anxiety in Patients Undergoing Third Molar Surgery
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dr. Damla Torul, Research Asistant, Ordu University
Other Study IDs: 2018-182
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: The control group consisted of patients who verbal explanation of the surgical procedure and the potential postoperative complications was given with a written informed consent document
  Interventions: Procedure: Third molar surgery
- Study group: Participants in the study group asked to watch impacted lower third molar extraction video which was previously uploaded to the internet with their own device. This video includes only visual components of the surgery such as anesthesia, incision, extraction and suturing. Patients in the second group were also informed verbally about the surgical procedure-possible postoperative complications and was given with a written informed consent document.
  Interventions: Procedure: Third molar surgery

INTERVENTIONS:
Procedure: Third molar surgery — Surgical extraction of impacted lower third molar tooth under local anesthesia

SUMMARY:
Third molar extraction is the most common surgical procedure in the field of oral and maxillofacial surgery and usually cause anxiety. Although different informed consent methods have been used previously, the most effective information method that provide the optimum anxiety management is still not clear. Therefore, investigators planned a clinical study to explore the effect of different information formats (verbal information with written document and verbal information with written document subsequent to watching video from internet) on peri-operative anxiety of the participants who scheduled to undergo impacted lower third molar surgery. Also, investigators aimed to explore the effect internet usage before the third molar surgery on the level of anxiety.

DETAILED DESCRIPTION:
The participants were randomly divided into two groups. The control group consisted of participants who informed verbally about the surgical procedure and the potential postoperative complications,. Also, a written informed consent document was given. Participants in the study group were asked to watch a video which was previously uploaded to the internet and was showed procedural details of an impacted right lower third molar extraction (with permission and written consent). Participants in the study group were also informed verbally about the surgical procedure-possible postoperative complications and was given with a written informed consent document. In both groups questions of the participants were answered by the same surgeon. To evaluate anxiety; participants were asked to complete 3 questionnaires one week before the procedure when taking appointment for surgery, just after watching video or informed verbally, immediately after the procedure and one week after the procedure.

ELIGIBILITY:
Inclusion Criteria:

patients;

* without systemic disease,
* have indication for third molar extraction,
* radiographic degree of impaction according to the classification of Winter (vertical and mesio-angular) and the classification of Pell and Gregory 2, or 3 and B

Exclusion Criteria:

patients who;

* has psychiatric illness and systemic disease,
* refused to watch the video,
* failed to fill out the forms for any reason,
* had incomplete data and wanted to withdraw from the study,
* had underwent a previous third molar surgery,
* had history of anxiety attacks and/or anxiolytic treatment,
* had unpleasant dental treatment experience could not cooperated,

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients who scheduled to underwent impacted lower third molar removal in the Oral and Maxillofacial Surgery Clinic of Ordu University between August 2018 to February 2019.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Anxiety change being assessed with Spielberger State Anxiety Inventory (STAI-S) | one week before the procedure when taking appointment for surgery, just after watching video or informed verbally, immediately after the procedure and one week after the procedure
  There are total 40 questions in STAI-S (20). For each question the patients score ranged from 1 (almost never) to 4 (almost always) points. The sum of the scores range from 20-80. The score between 36 to 41 refer the mean anxiety level, and the values above 41 classified as high level of anxiety.
Anxiety change being assessed with Modified Dental Anxiety Scale (MDAS) | one week before the procedure when taking appointment for surgery, just after watching video or informed verbally, immediately after the procedure and one week after the procedure
  MDAS consists of five questions in total which measures anxiety at different stages of dental treatment. 1 (no anxious) to 5 (very anxious) options are available for each question. The sum of the scores varies from 5 to 25 and the values between 19-25 indicates high dental anxiety.
Anxiety change being assessed with Amsterdam Preoperative Anxiety Inventory (APAIS) | one week before the procedure when taking appointment for surgery, just after watching video or informed verbally, immediately after the procedure and one week after the procedure
  APAIS is a scale consisting of 6 items, 3 of them are related to anesthesia and the others related to surgical procedure. The scoring ranges from 6 to 30 in total. The value of >11 is considered as high-anxiety level.
Trait Anxiety assessed with Spielberger Trait Anxiety Inventory (STAI-T) | one week before the procedure
  There are total 40 questions in d STAI-T (20). For each question the patients score ranged from 1 (almost never) to 4 (almost always) points. The sum of the scores range from 20-80. The score between 36 to 41 refer the mean anxiety level, and the values above 41 classified as high level of anxiety.

SECONDARY OUTCOMES:
Pain severity change | 1st, 3rd and 7th day after surgery
  Pain measured with Visual Analog scale (VAS) The pain levels of the patients were evaluated by a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (extremely pain).
Analgesic consumption per day | 1st, 3rd and 7th day after surgery
  Amount of analgesic consumption. High consumption show worse recovery

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet M Omezli, PhD, Study Director — Associate Professor
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results of the publication of the study
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: Contributors of the study will review requests